CLINICAL TRIAL: NCT00436800
Title: Gemcitabine and Oxaliplatin in First Line Metastatic or Recurrent Nasopharyngeal Carcinoma (NPC)
Brief Title: Gemcitabine and Oxaliplatin (GEMOX) in First Line Metastatic or Recurrent Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_9281
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-08

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Gemcitabine; Oxaliplatin

ARMS (1):
- 1 (Experimental): Gemcitabine on Day 1 followed by Oxaliplatin on Day 2. The regimen is given every 2 weeks to a maximum of 12 cycles.
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m² over 10mg/m²/min
Drug: Oxaliplatin — 100 mg/m² over 2 hours.

SUMMARY:
Primary objective:

To evaluate the response rate of biweekly gemcitabine and oxaliplatin (the GEMOX regimen) in the first line treatment of metastatic or recurrent nasopharyngeal carcinoma.

Secondary objectives:

To assess the toxicity, duration of response, time to progression, progression-free survival, overall survival and cancer-related symptoms in the first line treatment of patients with metastatic or recurrent NPC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically proven nasopharyngeal carcinoma (NPC) with metastatic or recurrent disease that is not amenable to potentially curative surgery or radiotherapy. They must not have prior chemotherapy for the treatment of metastatic or recurrent disease.
* Prior neoadjuvant, adjuvant or concurrent chemotherapy is allowed as long as a minimum period of 6 weeks has elapsed since the last day of treatment. This includes the use of carboplatin or cisplatin.
* Patients must have at least one uni-dimensional measurable lesion (according to RECIST criteria)
* Prior RT or surgery to the target lesion(s) is allowed as long as there is documented disease progression within the RT/ surgical field, and a minimum period of 6 weeks has elapsed since the last day of treatment.
* Eastern Cooperative Oncology Group performance status of 0-2
* No serious, uncontrolled medical conditions that may be aggravated by treatment.
* No other malignancy(s), except completely excised basal or squamous cell carcinoma of the skin, or completely treated carcinoma-in-situ of the cervix.
* Adequate hematological function:absolute granulocyte count > 1.5 x 10^9/L, platelet count > 100 x 10^9/L
* Adequate renal and hepatic functions:·serum creatinine < 1.25 x upper normal limit (UNL) or a calculated creatinine clearance > 50 mL/min·serum bilirubin < 2 x UNL and Aspartate aminotransferase/Alanine aminotransferase < 3 x UNL

Exclusion Criteria:

* Prior treatment with Oxaliplatin or Gemcitabine.
* Patients who have persistent grade 2 or more sensory and/or motor neuropathy, or ototoxicity resulting from prior cisplatin/ carboplatin.
* Active or past history of central nervous system metastasis from the primary tumor
* Potentially life-threatening infections
* Patients have used any investigational drug treatment in the month prior to inclusion.
* Pregnancy or not exercising appropriate birth control during the course of the study. Breast-feeding women

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Efficacy: Tumor response rate based on Response Evaluation Criteria in Solid Tumour (RECIST) criteria | Baseline to end of study
Safety: Clinical and laboratory criteria | Baseline to end of study
The incidence of adverse events based on National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 | Baseline to 30 days post treatment
Occurrence of serious adverse events (SAE) | Baseline to 30 days post treatment
Drop-out rate | End of study

SECONDARY OUTCOMES:
Toxicity, duration of response, time to progression, progression-free survival, overall survival and cancer-related symptoms. | Baseline to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Iris Chan, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong